CLINICAL TRIAL: NCT01032018
Title: Comparison of Depression Interventions After Acute Coronary Syndrome (CODIACS)
Brief Title: Comparison of Depression Interventions After Acute Coronary Syndrome
Acronym: CODIACS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of North Carolina, Chapel Hill (Other); Emory University (Other); Yale University (Other); Washington University School of Medicine (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Karina Davidson, Professor of Behavioral Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AAAE1932; RC2HL101663 (NIH)
Record Dates: First submitted 2009-12-11; First posted 2009-12-15 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-08

CONDITIONS: Acute Coronary Syndrome; Depression
Keywords: Acute coronary syndrome; Depression; Satisfaction with care
MeSH Terms: conditions — Acute Coronary Syndrome; Depression | interventions — Sertraline; Citalopram; Bupropion; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Referred Care (Active Comparator): Immediately after the initial post-ACS screening, the participant's physician will be notified in writing if the participant is depressed according to the BDI. Depending upon the physician's own evaluation of the participant, he or she may elect to defer depression treatment, initiate it, or to refer the patient to a mental health specialist.
  Interventions: Other: Standard care
- Stepped Care (Experimental): Stepped Care participants will be given a description of the choices available in this arm, including choosing antidepressant medication and/or telephone-based, Problem-Solving Therapy (PST). If the patient is randomized to Stepped Care, their physician will be informed that depression treatment is being provided by the trial. Patients will select their preferred treatment approach. Depression symptoms will be monitored to determine whether the patient is improving relative to his/her baseline score. Relapse monitoring and maintenance therapy will continue for the duration of the study.
  Interventions: Behavioral: Problem Solving Therapy; Drug: Sertraline, citalopram, or bupropion

INTERVENTIONS:
Behavioral: Problem Solving Therapy — Problem Solving Therapy (PST) will be administered by a trained provider. The concepts of PST will be taught to the participant in the first session and reinforced across subsequent sessions. Sessions will last between 30 and 60 minutes each and continue weekly for the duration of the study (6 months).
  Arms: Stepped Care
Drug: Sertraline, citalopram, or bupropion — Antidepressants should be started at the lowest dose, but should be adjusted upward to be within the therapeutic range within 1 week,with further adjustment higher in the therapeutic range possible at 3-4 weeks. Dosage of the first medication selected will be in the therapeutic range by 3 weeks of the initial step, as tolerated. If a patient cannot tolerate a particular treatment (i.e., intolerable side effects even with careful titration and clinical management), a switch to an alternative antidepressant or PST-PC after 2-4 weeks and 'restart' step 1.
  Sertraline: 25-150qam Citalopram: 10-40qam Bupropion: 100-450qam
  Arms: Stepped Care
Other: Standard care — Participants will receive standard of care from the current physicians
  Arms: Referred Care

SUMMARY:
Patients will be consented and screened within 2 to 6 months of the index ACS. Patients who have elevated depression (BDI>=15 or BDI>=10 assessed twice over two week period) and who continue to meet all of the trial's eligibility criteria will be consented. Through informed consent, both arms of the trial will be described with equipoise as to these approaches to postACS depression care. Patients who consent to randomization will be enrolled in the treatment trial.

The intervention phase will be 6 months, and hence the final outcome assessments will be performed approximately 9 months after the index ACS. Interim measures of depression will be obtained at 2 and 4 months post-enrollment. Major adverse cardiac events and all-cause mortality will also be ascertained at 6 months post-enrollment. Quality assurance by an independent medical event adjudication committee using prospective guidelines will be employed.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized for ACS defined as unstable angina or MI
* BDI greater or equal to 10 and < 15 2-6 months post-ACS on each of 2 occasions, or BDI greater than 15 on one occasion
* Age at least 35 years
* Fluent in English or Spanish
* Able to complete baseline assessment within 2-6 months of index ACS event
* Able and willing to provide informed consent

Exclusion Criteria:

* Presence of non-cardiac condition likely to terminate fatally within 1 year
* Inaccessibility for intervention or follow-up (e.g., plans to move from the area)
* Cognitive impairment
* Need for immediate psychiatric intervention (i.e., requiring hospitalization or psychiatric intervention within 72 hours)
* Suicidal ideation
* Major psychiatric co-morbidity (current or by history) including active psychosis, bipolar disorder, or overt personality disorder
* Active substance abuse or dependency
* Chronic renal failure (receiving chronic dialysis treatment, or estimated glomerular filtration rate"…[eGFR] < 30 ml/min/1.73 m2) or moderate/severe liver disease (e.g., esophageal varices, portal hypertension, encephalopathy, GI bleeding)
* Participation in another clinical trial for the treatment of depression.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karina W Davidson, PhD, Principal Investigator — Columbia University; J Thomas Bigger, MD, Principal Investigator — Columbia University; Robert Carney, PhD, Principal Investigator — Washington University School of Medicine; Kenneth Freedland, PhD, Principal Investigator — Washington University School of Medicine
Locations (5):
- United States (5):
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Washington University, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Trustees of the University of Pennsylvania, Penn Cardiac Center at Mercer Bucks, Yardley, Pennsylvania

REFERENCES:
- [Result] Davidson KW, Bigger JT, Burg MM, Carney RM, Chaplin WF, Czajkowski S, Dornelas E, Duer-Hefele J, Frasure-Smith N, Freedland KE, Haas DC, Jaffe AS, Ladapo JA, Lesperance F, Medina V, Newman JD, Osorio GA, Parsons F, Schwartz JE, Shaffer JA, Shapiro PA, Sheps DS, Vaccarino V, Whang W, Ye S. Centralized, stepped, patient preference-based treatment for patients with post-acute coronary syndrome depression: CODIACS vanguard randomized controlled trial. JAMA Intern Med. 2013 Jun 10;173(11):997-1004. doi: 10.1001/jamainternmed.2013.915. PMID 23471421
- See also: Related Info — http://www.nhlbi.nih.gov/
- See also: Baseline design paper — http://dx.doi.org/10.1016/j.cct.2012.05.005

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from sites connected with 5 field centers from March 18, 2010, to January 9, 2012. To be eligible, participants had to demonstrate elevated depressive symptoms on the BDI 2 to 6 months after hospitalization for an ACS.
Pre-assignment Details: 724 patients were medically eligible for participation in the study, of which 150 consented to randomization and were enrolled.
Groups:
- Referred Care: The participant's primary care provider was notified in writing of the finding of elevated depressive symptoms and encouraged to implement a provider-preferred depression treatment. Depending on the provider's evaluation of the participant, he or she elected to defer depression treatment, to initiate it, or to refer the participant to a mental health specialist.
- Stepped Care: The participant had a choice of Problem Solving Therapy (PST), pharmacotherapy, a combination of the two, or neither. The participant had a 15-minute information session on the benefits of drawbacks of each type of therapy and medication, after which the preferred treatment was chosen.
Period: Overall Study
Arm/Group | Referred Care | Stepped Care
Started | 77 | 73
Completed | 71 | 67
Not Completed | 6 | 6
Not completed — Lost to Follow-up | 6 | 5
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Referred Care | Stepped Care | Total
Number analyzed (Participants) | 77 | 73 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (11.1) | 59.2 (9.7) | 59.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 30 | 63
  Male | 44 | 43 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 16 | 29
  Not Hispanic or Latino | 64 | 56 | 120
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 27 | 23 | 50
  White | 42 | 42 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 7 | 14
Beck Depression Inventory Score, continuous [Mean (Standard Deviation); unit: Scores on a scale] — The Beck Depression Inventory (BDI) is a 21-item multiple choice, self-report instrument that is used to assess the severity of symptoms of depression. The score ranges from 0 (no symptoms) to 63 (worst symptoms).
  Scores on a scale | 20.6 (7.8) | 21.0 (7.6) | 20.8 (7.7)
Beck Depression Inventory Score, categorical [Number; unit: participants]
  BDI score < 16 | 27 | 21 | 48
  BDI score >= 16 | 50 | 52 | 102
Type of presenting acute coronary syndrome [Number; unit: participants] — MI = Myocardial Infarction
  participants
    Unstable angina | 35 | 35 | 70
    Non-ST segment elevated MI | 19 | 18 | 37
    ST-segment elevated MI | 21 | 19 | 40
    Bundle branch block/uncertain type of MI | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptom Reduction
Description: Symptoms of depression were assessed using the Beck Depression Inventory (BDI). This 21-question, multiple choice self-report instrument includes items pertaining to symptoms of depression, including hopelessness and irritability, physical symptoms such as fatigue, and thoughts such as guilt. Each item has at a set of four possible responses, ranging in intensity for least intense to most intense. The total score is calculated by adding the responses to each item. Higher scores indicate more severe depressive symptoms. The total score on the scale ranges from 0 to 63. Total scores on the scale of less 10 indicate minimal depression; total scores between 10 and 15 indicate mild depression; and total scores greater than 16 indicate a probable clinical diagnosis of depression.
Time Frame: Change from depression at baseline to depression at 6-months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Referred Care | Stepped Care
Number analyzed (Participants) | 77 | 73
Scores on a scale | -6.6 (1.0) [-8.5 to -4.8] | -10.1 (0.9) [-12.0 to -8.1]
Statistical Analysis 1: Comparison: Referred Care vs Stepped Care; The trial was powered to detect a between-group difference in the 6-month change in depression symptoms. Assuming 5% attrition rate, we estimated that a sample of 150 patients would be needed to have 80% power to detect a clinically meaningful differential change in depression scores between groups of 0.46 SD; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis; Difference of back-transformed means. = -3.5, 95% CI [-6.1 to -0.7]

2. Primary Outcome: Cost for Healthcare Utilization (Psychiatric Medications, Hospitalizations, Cardiac Procedures, Outpatient Services)
Time Frame: 6 months after randomization
Measure: Mean (Standard Error); unit: dollars
Arm/Group | Referred Care | Stepped Care
Number analyzed (Participants) | 77 | 73
dollars | 4289.23 (826.56) | 4358.02 (883.76)

ADVERSE EVENTS:
Time Frame: 2, 4, and 6 months after enrollment
Arm/Group | Referred Care | Stepped Care
Serious Adverse Events (participants affected / at risk) | 8/77 | 7/73
Other Adverse Events (participants affected / at risk) | 63/77 | 59/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Referred Care (N=77) | Stepped Care (N=73)
Death (General disorders) | 0 | 1
GI bleeding (Gastrointestinal disorders) | 1 | 2
MRSA Infection (Infections and infestations) | 1 | 0
Internal bleeding (Blood and lymphatic system disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 3
Stroke (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Referred Care (N=77) | Stepped Care (N=73)
Abdominal hernia (Injury, poisoning and procedural complications) | 0 | 1
Worsened agitation (Psychiatric disorders) | 7 | 4
Anemia (Blood and lymphatic system disorders) | 0 | 1
Worsened anxiety/nervousness (Psychiatric disorders) | 5 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Blood in stool (Gastrointestinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Worsened decreased appetite (Gastrointestinal disorders) | 8 | 6
Worsened diarrhea (Gastrointestinal disorders) | 3 | 5
Diverticulitis (Gastrointestinal disorders) | 1 | 0
Worsened dizziness (Nervous system disorders) | 0 | 1
Worsened drowsiness (Nervous system disorders) | 7 | 2
Worsened dry mouth (Skin and subcutaneous tissue disorders) | 14 | 8
Dysgeusia (Nervous system disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Ear bleeding (Ear and labyrinth disorders) | 0 | 1
Fall (Musculoskeletal and connective tissue disorders) | 2 | 1
GI problems (Gastrointestinal disorders) | 25 | 30
Gum bleeding (Blood and lymphatic system disorders) | 1 | 2
Headaches (Nervous system disorders) | 0 | 2
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 1
Hip pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Worsened increase in appetite (Gastrointestinal disorders) | 5 | 9
Worsened indigestion (Gastrointestinal disorders) | 15 | 14
Worsened insomnia (Nervous system disorders) | 3 | 4
Irregular menstrual period (Gastrointestinal disorders) | 1 | 0
Joint pains (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Knee injury (Musculoskeletal and connective tissue disorders) | 0 | 1
Leg edema (Cardiac disorders) | 22 | 15
Low potassium (Metabolism and nutrition disorders) | 0 | 1
Middle ear effusion (Ear and labyrinth disorders) | 0 | 1
Mood disturbance (Psychiatric disorders) | 1 | 0
Worsened nausea (Gastrointestinal disorders) | 8 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Nosebleed (Blood and lymphatic system disorders) | 2 | 7
Numbness of arms and legs (Nervous system disorders) | 1 | 1
Oral bleedin (Blood and lymphatic system disorders) | 1 | 0
Pain (Nervous system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Pruritus (Nervous system disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rectal bleeding (Gastrointestinal disorders) | 4 | 5
Worsened sexual side effects (Reproductive system and breast disorders) | 5 | 3
Strep throat (Infections and infestations) | 0 | 1
Worsened sweating (Metabolism and nutrition disorders) | 4 | 6
Tingling of fingers and toes (Nervous system disorders) | 1 | 0
Worsened tremors (Nervous system disorders) | 6 | 3
Upper respiratory infection (Infections and infestations) | 1 | 0
Upset stomach (Gastrointestinal disorders) | 33 | 35
Urinary tract infection (Infections and infestations) | 0 | 2
Vaginal bleeding (Reproductive system and breast disorders) | 1 | 0
Varicose veins (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes